CLINICAL TRIAL: NCT03100526
Title: Patient Aligned Care Team (PACT) Intensive Management (PIM) Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veteran Affairs Office of Patient Care Services (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PIM Evaluation
Record Dates: First submitted 2017-02-10; First posted 2017-04-04 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Primary Health Care; Health Care Costs
Keywords: High-Risk Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention--PACT Intensive Management (Experimental): The intervention is the PACT Intensive Management Program (PIM) which provides intensive interdisciplinary care planning, care coordination, patient self-management support, and tailored goal setting based on patient needs and preferences, and additional care management services.
  Interventions: Behavioral: PACT Intensive Management
- Usual care (No Intervention): High-Risk patients receiving care in PACT.

INTERVENTIONS:
Behavioral: PACT Intensive Management — Purpose: Implement a Patient Aligned Care Team (PACT) model that identifies and proactively manages Veterans at the highest risk for hospital admission and death while they are still in the ambulatory care setting.
  Goal:
  * Reduce emergency department and urgent care utilization, hospitalization, and mortality in complex, high risk patients
  * Improve Veteran and staff satisfaction
  Objectives:
  * Maintain the patient in the home setting as much as possible
  * Secure appropriate home environment to facilitate health and well-being
  * Utilize comprehensive team-based care
  * Engage appropriate VHA programs to provide interdisciplinary, coordinated, and timely management of complex medical issues
  Other Names: PIM
  Arms: Intervention--PACT Intensive Management

SUMMARY:
Purpose: Implement a Patient Aligned Care Team (PACT) model that identifies and proactively manages Veterans at the highest risk for hospital admission and death while the patient is still in the ambulatory care setting.

Goal:

* Reduce emergency department and urgent care utilization, hospitalization, and mortality in complex, high risk patients
* Improve Veteran and staff satisfaction

Objectives:

* Maintain the patient in the home setting as much as possible
* Secure appropriate home environment to facilitate health and well-being
* Utilize comprehensive team-based care
* Engage appropriate Veteran Health Administration (VHA) programs to provide interdisciplinary, coordinated, and timely management of complex medical issues

ELIGIBILITY:
Inclusion Criteria:

* selected for intensive management

Exclusion Criteria:

* enrolled in other intensive case management at VA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2210 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
VA health care cost | 2 years (two 1-year points)
  Total costs of VA care, including inpatient, outpatient, pharmacy and fee-basis services.

SECONDARY OUTCOMES:
Healthcare Utilization | 2 years (two 1-year points)
  VA central repository administrative data will be analyzed to calculate utilization of hospital, emergency and outpatient primary and specialty care. This information will be electronically abstracted through the VA central repository administrative data center
Total Medicare Cost | 2 years (two 1-year points)
  Data will be extracted from VHA's Corporate Data Warehouse to capture patient Medicare cost. Medicare claims data to measure total patient inpatient and outpatient cost for services reimbursed by Medicare. Inpatient cost will be measured as cost for total acute hospitalizations, and subcategories: medical, surgical, psychiatric, rehabilitation, hospice and ambulatory care-sensitive conditions. Outpatient cost will be measured as the cost for combined visits in VHA and elsewhere reimbursed by Medicare in 9 categories: primary care, specialty care, mental health, surgical, home health, nursing home, diagnostic, rehabilitation and ED.
Total Medicare Utilization | 2 years (two 1-year points)
  Data will be extracted from VHA's Corporate Data Warehouse to capture patient utilization. Medicare claims data to measure total patient inpatient and outpatient utilization for services reimbursed by Medicare. Inpatient utilization will be measured as counts of total acute hospitalizations, and subcategories: medical, surgical, psychiatric, rehabilitation, hospice and ambulatory care-sensitive conditions. Outpatient utilization will be measured as the number of combined visits in VHA and elsewhere reimbursed by Medicare in 9 categories: primary care, specialty care, mental health, surgical, home health, nursing home, diagnostic, rehabilitation and ED.

OTHER OUTCOMES:
Patient Engagement | 2 years (two 1-year points)
  The investigators will look at patient PIM enrollment data by utilizing qualitative data. The data will be collected through qualitative interviews with patients and PACT providers.
  Provider Interviews questions:
  Tell me what kinds of things you and your team have been doing to try to engage patients What types of patients have you been able to engage most successfully? Once patients have started to engage with the PIM team, how do you prioritize what to work on with them?
  Patient Interview questions:
  Has working with the PIM team made a difference in your health? Have you changed how you take care of yourself since you have been part of PIM? If you were going to tell another Veteran about this program, what would you say (are the pros and cons)? How would you say you have benefitted from being in this program? What have been the drawbacks of being in this program?
Functional status | 2 years (two 1-year points)
  Patient report of their physical, social, and mental functional status is routinely collected as part of their medical visit as health factor data. The data will be abstracted through the VA central repository administrative data. The variables used to measure functional status are the following:
  * In general, how would you rate your satisfaction with your social activities and relationships? (Excellent, Very good, Good, Fair, Poor)
  * In general, please rate how well you carry out your usual social activities and roles. (This includes activities at home, at work and in your community, and responsibilities as a parent, child, spouse, employee, friend, etc.) (Excellent, Very good, Good, Fair, Poor)
  * Administer Katz Index of Independence in Activities of Daily Living (Independence=1 point; dependence = 0 points for each of the six item pairs)
  * Administer the Lawton Instrumental Activities of Daily Living (IADL) Scale (score 0-8)
Patient Quality of Life Status | 2 years (two 1-year points)
  Patient assessment of their quality of life collected as part of their medical care as a health factor. This information will be electronically abstracted through the VA central repository administrative data center. The variables used to assess a patient's quality of life are the following:
  * Patient's self-rating of quality of life in general: Excellent, Very Good, Good, Fair, Poor
  * Patient's self-rating of mental health, including mood and ability to think: Excellent, Very Good, Good, Fair, Poor
Patient Symptom Burden | 2 years (two 1-year points)
  Patient assessment of symptom burden is routinely collected as part of their care and documented in their medical record and will be electronically abstracted through the VA central repository administrative data center. Mental Health and physical burdens are abstracted from the medical record utilizing ICD-9 and ICD-10 code. It will be assessed as yes/no if present.
Anxiety | 2 years (two 1-year points)
  Generalized Anxiety Disorder 2-item (GAD-2): (Not at all; several days; More than half the days, nearly every day). The higher the score the higher the anxiety.
Substance Abuse | 2 years (two 1-year points)
  The 3-item AUDIT-C scored on a scale of 0-12; Drugs: How many times in the past year, have you used an illegal drug or used a prescription medication for nonmedical reasons? (Yes/No, Number of times). The greater the score the worse the substance abuse status.
Cognitive Status | 2 years (two 1-year points)
  The Blessed-Short and/or the Mini-Cog where the lower the score the more impairment.
Pain level | 2 years (two 1-year points)
  Pain in past 24 hours on scale of 0 = no pain, to 10 = worst pain imaginable.
Shortness of Breath | 2 years (two 1-year points)
  Shortness of breath in past 24 hours on a scale of 0, no shortness of breath, to 10, worst imaginable.
Problems with constipation | 2 years (two 1-year points)
  Constipation in past 24 hours on a scale from 0, no constipation, to 10, worst imaginable.
Sleep Problems | 2 years (two 1-year points)
  Sleep problems in past 24 hours on a scale from 0, no sleep problems, to 10, worst imaginable.
Level of Fatigue | 2 years (two 1-year points)
  Fatigue in past 24 hours on a scale from 0, no fatigue, to 10, worst imaginable.
Risk of Falls | 2 years (two 1-year points)
  Falls (Patient reports no falls in past 12 months;Patient reports no problems with walking or balance; Patient reports problems with walking or balance; Patients reports falls in past 12 months
Implementation Outcome/challenges | 2 years (two 1-year points)
  Implementation barriers and facilitators, feasibility, and sustainability will be obtained through stakeholder interviews of patients, staff and facility leaders. PIM Staff topics include program goals, patient enrollment, engagement strategies, patient decision making; target population, gaps in care, care coordination, readiness, resource adequacy, and sustainability. PIM program leader topics include lessons learned, impact and sustainability, and implementation process. Patient topics include experience in program, engagement in care and suggestions for improvement. PACT teamlet topics include exposure to PIM, the impact on workload, the services PIM provides, feasibility of providing PIM services, impact and sustainability of PACT on working with PIM team. Facility leaders topics include PIM program goals, specialty service programs, target population, and services for high-risk patients, PACT functioning, PIM affects patients on services, and facility.
Primary Care Staff Job Satisfaction | 3 years (two waves)
  We will survey Primary Care Providers (PCPs) (physicians, MDs/DOs; nurse practitioners, NPs; physician assistants, PAs) and nurses (registered nurses, RNs; licensed practical nurses, LPNs; licensed vocational nurses-LVNs) at the five healthcare systems that have a PIM team. We will use both online using RedCap and paper-and-pen versions of the survey to increase response rate. We will survey Primary Care staff at baseline and one year later. Primary Care Staff Job Satisfaction is measured by a single item "Overall, I am satisfied with my job," rated on a 5-point Likert agreement scale. (Strongly disagree, Disagree, Neither agree nor disagree, Agree, Strongly agree). The higher the score the higher the satisfaction.
  • Overall, I am satisfied with my job. (Strongly disagree, Disagree, Neither agree nor disagree, Agree, Strongly agree). The higher the score the higher the satisfaction.
Primary Care staff Intention to Stay at the VA | 3 years (two waves)
  We will survey Primary Care Providers (PCPs) (physicians, MDs/DOs; nurse practitioners, NPs; physician assistants, PAs) and nurses (registered nurses, RNs; licensed practical nurses, LPNs; licensed vocational nurses-LVNs) at the five healthcare systems that have a PIM team. We will use both online using RedCap and paper-and-pen versions of the survey to increase response rate. We will survey Primary Care staff at baseline and one year later. Intention to Stay at the VA is measured by a single item "I intend to continue working in PC at the VA for the next two years," rated on a 5-point Likert agreement scale. (Strongly disagree, Disagree, Neither agree nor disagree, Agree, Strongly agree). The higher the score the higher the satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Rubenstein, MD, Principal Investigator — VAGLAHS- WLA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon J, Chang E, Rubenstein LV, Park A, Zulman DM, Stockdale S, Ong MK, Atkins D, Schectman G, Asch SM. Impact of Primary Care Intensive Management on High-Risk Veterans' Costs and Utilization: A Randomized Quality Improvement Trial. Ann Intern Med. 2018 Jun 19;168(12):846-854. doi: 10.7326/M17-3039. Epub 2018 Jun 5. PMID 29868706
- [Derived] Chang ET, Zulman DM, Asch SM, Stockdale SE, Yoon J, Ong MK, Lee M, Simon A, Atkins D, Schectman G, Kirsh SR, Rubenstein LV; PIM Executive Committee and Demonstration Sites. An operations-partnered evaluation of care redesign for high-risk patients in the Veterans Health Administration (VHA): Study protocol for the PACT Intensive Management (PIM) randomized quality improvement evaluation. Contemp Clin Trials. 2018 Jun;69:65-75. doi: 10.1016/j.cct.2018.04.008. Epub 2018 Apr 23. PMID 29698772

DOCUMENTS (1):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT03100526/Prot_001.pdf